CLINICAL TRIAL: NCT02614222
Title: Computer Assisted Instrument Guidance (CAIG) For Orthopedic Peripheral Nerve Blocks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clear Guide Medical (Industry)
Collaborators: The Cooper Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CGM 15-002
Record Dates: First submitted 2015-11-19; First posted 2015-11-25 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-06

CONDITIONS: Peripheral Nerve Blocks
Keywords: Computer Assisted Instrument Guidance (CAIG); Peripheral Nerve Block; Clear Guide ONE; Needle path; Needle Guidance; Ultrasound

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peripheral Nerve Block with CAIG (Experimental): The participants in this group (test group) will utilize the same procedure utilizing existing ultrasound equipment with the supplemental CAIG system.
  Interventions: Device: Peripheral Nerve Blocks with CAIG
- Peripheral Nerve Block without CAIG (No Intervention): The participants in the control group will receive the procedure with traditional ultrasound methods and equipment.

INTERVENTIONS:
Device: Peripheral Nerve Blocks with CAIG — The Clear Guide ONE is a Computer Assisted Instrument Guidance (CAIG) device which supplements existing ultrasound capabilities. The participants randomly selected (out of 100 patients) for use of the Clear Guide ONE (test group) will receive ultrasound guidance as well as CAIG from the MDs performing the procedure.
  Other Names: Clear Guide ONE
  Arms: Peripheral Nerve Block with CAIG

SUMMARY:
The objective of this research is to determine if the addition of the Clear Guide ONE, a Computer Assisted Instrument Guidance (CAIG) system, provides improvement over existing ultrasound guided, needle-based procedures for peripheral nerve blocks. The ultrasound can visualize the targeted vessel or nerve, but the addition of the CAIG may help the clinician better guide the needle to the target.

DETAILED DESCRIPTION:
This pilot study will be a randomized, single-blinded control trial. The clinicians cannot be blinded, but the person questioning the patient post-op to determine success rate will be blinded. There will be two randomized groups of patients: control and test. The control group will receive the procedure with traditional methods and equipment currently in use at Cooper University. The test group will receive the same procedure utilizing existing ultrasound equipment with the supplemental CAIG system.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing orthopedic surgery who are candidates for peripheral nerve blocks for control of postoperative pain
* Able to give written informed consent

Exclusion Criteria:

* Unable to give informed consent
* Patients in whom regional anesthesia is contradicted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-10-26; Primary Completion 2016-05-25 (Actual); Study Completion 2016-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronak Desai, DO, Principal Investigator — The Cooper Health System
Locations (1):
- The Cooper Health System, Camden, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Peripheral Nerve Block With CAIG | Peripheral Nerve Block Without CAIG
Started | 13 | 14
Completed | 13 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peripheral Nerve Block With CAIG | Peripheral Nerve Block Without CAIG | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 19
  >=65 years | 3 | 5 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  United States | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Time Needed to Correctly Identify the Neural Structure(s) and Induce the Peripheral Nerve Block
Time Frame: Immediately after intervention (within 2 hours)
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Peripheral Nerve Block With CAIG | Peripheral Nerve Block Without CAIG
Number analyzed (Participants) | 13 | 14
Minutes | 2.606944444 (1.445017966) | 2.179761905 (0.510579467)

2. Secondary Outcome: Clinician Rating of the Device
Description: Clinician rates the device on a scale of 1-10. This also includes a questionnaire.
Time Frame: Immediately following intervention (within 2 hours)
Population: Data for this outcome measure was not collected
Arm/Group | Peripheral Nerve Block With CAIG | Peripheral Nerve Block Without CAIG
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Attempts
Description: Number of instrument pricks before target is reached
Time Frame: Immediately following intervention (within 2 hours)
Population: This data was not collected for 3 (out of 27) participants.
Measure: Mean (Standard Deviation); unit: Attempts
Arm/Group | Peripheral Nerve Block With CAIG | Peripheral Nerve Block Without CAIG
Number analyzed (Participants) | 12 | 12
Attempts | 1 (0) | 1 (0)

4. Secondary Outcome: Number of Times Needle Needs Repositioning
Time Frame: Immediately following intervention (within 2 hours)
Population: Data for this outcome measure was not collected.
Arm/Group | Peripheral Nerve Block With CAIG | Peripheral Nerve Block Without CAIG
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Patient Satisfaction Recorded on Post-op Day 1 Using Questionnaire
Description: Patient satisfaction will be recorded in the hospital or via phone on post-op day 1, on a 10-point scale (10 being most satisfied), using a questionnaire.
Time Frame: Post-op day 1
Population: This data was not collected for 5 (out of 27) participants.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Peripheral Nerve Block With CAIG | Peripheral Nerve Block Without CAIG
Number analyzed (Participants) | 10 | 12
Units on a Scale | 8.727272727 (1.489356176) | 9.181818182 (1.662418829)

6. Secondary Outcome: Number of Patients That Needed Rescue Opioids
Time Frame: During hospital stay (maximum 3 days)
Population: This data was not collected for 4 (out of 27) patients
Measure: Count of Participants; unit: Participants
Arm/Group | Peripheral Nerve Block With CAIG | Peripheral Nerve Block Without CAIG
Number analyzed (Participants) | 12 | 11
Participants | 6 | 5

7. Secondary Outcome: Incidence of Postoperative Nausea and Vomiting
Description: Number of participants that reported postoperative nausea and vomiting
Time Frame: During hospital stay (maximum 3 days)
Population: This data was not collected for 4 (out of 27) participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Peripheral Nerve Block With CAIG | Peripheral Nerve Block Without CAIG
Number analyzed (Participants) | 11 | 12
Participants | 0 | 2

8. Secondary Outcome: Undesired Muscle Weakness Measured Subjectively
Description: Number of participants that report undesired muscle weakness. Undesired muscle weakness will be measured subjectively - whether patient unable to ambulate and/or requiring the use of an immobilizer.
Time Frame: During hospital stay (maximum 3 days)
Population: This data was not collected for 6 (out of 27) participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Peripheral Nerve Block With CAIG | Peripheral Nerve Block Without CAIG
Number analyzed (Participants) | 11 | 10
Participants | 2 | 1

ADVERSE EVENTS:
Arm/Group | Peripheral Nerve Block With CAIG | Peripheral Nerve Block Without CAIG
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 0/13 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No